CLINICAL TRIAL: NCT06847087
Title: Study of the Adequacy Between Calcium Supplementation and Dietary Intake in Treatment-naive Patients After Fracture With a Fracture Suspected of Being Due to Bone Insufficiency, Consulting a Rheumatologist for the First Time in at Least 5 Years.
Brief Title: Study of the Adequacy Between Calcium Supplementation and Dietary Intake in Treatment-naive Patients After a Fracture
Acronym: MONTE-CRIST'OS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier de Colmar (Other)
Responsible Party: Sponsor
Other Study IDs: HCC-008; ID-RCB 2024-A02648-39 (Other: Hôpitaux Civils de Colmar)
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Osteoporosis, Post-Traumatic; Calcium Supplementation; Osteoporosis, Management Care, Fracture
MeSH Terms: conditions — Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Self-questionnaire — Assessment of the inadequacy between dietary and medicinal calcium intake by the Fardellone self-questionnaire and the patient's clinical record

SUMMARY:
Osteoporosis is a disease that causes many fractures. However, treatments exist such as anti-osteoporotic treatments, vitamin D supplementation and an adaptation of calcium intake. 80% of patients with an indication for anti-osteoporotic treatment are never treated with these anti-osteoporotic treatments after a first fracture. On the other hand, more than 84% of them are supplemented with calcium and vitamin D. It often appears in the practice of rheumatologists that some patients are supplemented while their dietary intake is sufficient, and vice versa. The objective of the study is therefore to take stock of the (in)adequacy between the dietary intake of patients and the supplementation prescribed to them following an osteoporotic-like fracture.

ELIGIBILITY:
Inclusion Criteria:

* Patient meeting a first rheumatologist after a fracture suspected of being due to bone insufficiency, whether or not he is already treated for osteoporosis
* Age ≥ 18 years
* Patient followed in one of the three investigation centers within the framework of the bone sector.
* Patient affiliated to a social security system

Exclusion Criteria:

* Patient refusing to participate in the study
* Patient already followed by a rheumatologist
* Legal incapacity or any physical, psychological, social or geographical condition likely to hinder the patient's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting in a rheumatology department for a hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients deficient, within the norm and above the norm with or without supplementation | Day 1
  percentage of patients

SECONDARY OUTCOMES:
Previously performed bone densitometry | Day 1
  Results of densitormetry by a T score
Prevalence of a history of fracture | Day 1
  Number of bone fractures the patient has already had before inclusion
First indication for the initiation of anti-osteoporotic treatment. | Day 1
  Date of the first indication for the initiation of an anti-osteoporotic treatment.
  This date is appearing in the medical record
Duration without treatment before a fracture occurs | Day 1
  Duration without treatment before a fracture occurs and type of the treatment
Number of participants who need for readjustment by the rheumatologist after inclusion | Day 1
  Implementation of educational measures by the rheumatologist in the event of inadequacy and optimization of anti-osteoporotic treatments

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Civils de Colmar, Colmar, France